CLINICAL TRIAL: NCT06123338
Title: A Single-Arm, Multicenter Phase 2 Study of Neoadjuvant Pembrolizumab With Trastuzumab and Chemotherapy in Resectable HER2+ Esophagogastric Tumors
Brief Title: A Study of Pembrolizumab With Trastuzumab and Chemotherapy in People With Esophagogastric Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-124
Record Dates: First submitted 2023-11-03; First posted 2023-11-08 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Esophageal Cancer; Gastric Adenocarcinoma; HER2 Gene Mutation
Keywords: HER2+ Esophageal cancer; Esophageal Cancer; Gastric Adenocarcinoma; HER2+ GEJ cancer; HER2 IHC3+ expression; IHC 2+/FISH>2.0 expression; Esophagogastric cancer; Memorial Sloan Kettering Cancer Center; 23-124
MeSH Terms: conditions — Esophageal Neoplasms | interventions — pembrolizumab; Trastuzumab; Oxaliplatin; Capecitabine; Fluorouracil; Docetaxel

STUDY DESIGN:
Intervention Model Description: This is a single-arm phase 2 study in which patients with resectable HER2-positive EGC will receive peri-operative trastuzumab and pembrolizumab in combination with chemotherapy.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Esophagogastric Cancer (Experimental): Participants will have a diagnosis of resectable HER2+ (IHC 3+ or IHC 2+/FISH ratio >2.0) esophageal, GEJ or gastric cancer.
  Interventions: Drug: Pembrolizumab; Drug: Trastuzumab; Drug: Oxaliplatin; Drug: Capecitabine; Drug: 5-Fluorouracil; Drug: Docetaxel

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab will be administered on an every 3-week dosing schedule
Drug: Trastuzumab — Trastuzumab will be administered on an every 3-week dosing schedule
Drug: Oxaliplatin — Oxaliplatin every 3 weeks, +/-7 days
Drug: Capecitabine — Capecitabine twice daily on days 1 to 14 every 3 weeks or 5-FU on days 1 to 5 every 3 weeks
Drug: 5-Fluorouracil — 5-Fluorouracil administered as a 24 hour IV continuous infusion once every 2 weeks
Drug: Docetaxel — Docetaxel administered intravenously once every 2 weeks.

SUMMARY:
The purpose of this study to find out whether adding trastuzumab and pembrolizumab to standard chemotherapy is an effective treatment for resectable HER2+ esophagogastric cancer.

DETAILED DESCRIPTION:
Eligible patients will receive 8 peri-operative cycles of pembrolizumab and trastuzumab with chemotherapy (fluoropyrimidine/oxaliplatin doublet for patients initially enrolled and subsequently FLOT [5-fluorouracil, oxaliplatin and docetaxel] followed by pembrolizumab and trastuzumab maintenance to complete 1 total year of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older at time of signing informed consent.
* ECOG performance status 0-1.
* HER2+ esophageal, GEJ, or gastric adenocarcinoma biopsy or resection specimen as defined by local HER2 IHC3+ or IHC 2+/FISH>2.0 expression.
* Complete surgical resection of the primary tumor must be achievable
* Demonstrate adequate organ function as defined in Table 1.

Table 1 - Organ Function Requirements for Eligibility Hematological

* Absolute neutrophil count (ANC): ≥1,500 /mcL
* Platelets: ≥100,000 / mcL
* Hemoglobin: ≥8 g/dL Renal
* Creatinine clearance: ≥ 50 mL/minute Hepatic
* Serum total bilirubin: ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN. Except patients with Gilbert's disease (≤3x ULN)
* AST and ALT: ≤ 2.5 X ULN
* Albumin: >3 mg/dL Coagulation
* International normalized ratio (INR) OR prothrombin time (PT) Activated partial thromboplastin time (aPTT): <1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
* Male participants: A male participant must agree to use contraception as detailed in Section 15.3 of this protocol during the treatment period and for at least 230 days (5 terminal half-lives of trastuzumab [140] plus an additional 90 days [spermatogenesis cycle]) after the last dose of study treatment and refrain from donating sperm during this period.
* Female participants: A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  1. Not a woman of childbearing potential (WOCBP) as defined in section 15.3 OR
  2. A WOCBP who agrees to follow the contraceptive guidance in section 15.3 during the treatment period and for at least 170 days (140 days plus an additional 30 days [menstruation cycle]) after the last dose of study treatment.

Exclusion Criteria:

* Presence of metastatic or recurrent disease.
* Has received prior treatment for esophagogastric cancer
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-CTLA-4 agent.
* Has received prior therapy with an anti-HER2 agent
* Left ventricular ejection fraction <50% within 1 month of screening by MUGA or echocardiogram. Patients with an ejection fraction 45-49% may be permissible in the absence of any cardiac symptoms, if cleared by a cardiologist, and per the investigator's discresion.
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Patients who have received acute, low dose, systemic immunosuppressant medications (e.g., dexamethasone containing antiemetic regimen or steroids as CT scan contrast premedication) may be enrolled.
* The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed.
* Has a known history of active TB (Bacillus tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients
* Has been diagnosed or treated for another malignancy in the past 3 years (not including non-melanoma skin cancer)
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* A WOCBP who has a positive urine pregnancy test within 72 hours prior to allocation. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Has had an allogeneic tissue or solid organ transplant
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease; systemic lupus erythematosus; Wegener syndrome [granulomatosis with polyangiitis]; myasthenia gravis; Graves' disease; rheumatoid arthritis, hypophysitis, uveitis) within the past 3 years prior to the start of treatment. The following are exceptions to this criterion:

  * Subjects with vitiligo or alopecia
  * Subjects with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement or psoriasis not requiring systemic treatment.
  * Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* Is unwilling to give written informed consent, unwilling to participate, or unable to comply with the protocol for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | 2 years
  EFS is defined as the time from start of treatment to time of disease progression, recurrence, or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Yelena Janjigian, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (10):
- United States (10):
  - Massachusetts General Hospital (Data Collection Only), Boston, Massachusetts
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (Limited protocol activity), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York
  - University of Pennsylvania (Data Collection Only), Philadelphia, Pennsylvania
  - MD Anderson Cancer Center (Data Collection Only), Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org